CLINICAL TRIAL: NCT00755287
Title: A Multicenter, Randomized, Open-label, Active-controlled Study to Compare the Safety, Tolerability and Effect on Glycemic Control of Taspoglutide Versus Insulin Glargine in Insulin-naïve Type 2 Diabetic Patients Inadequately Controlled With Metformin and Sulphonylurea Combination Therapy
Brief Title: A Study of the Safety, Tolerability and Effect on Glycemic Control of Taspoglutide Versus Insulin Glargine in Insulin Naive Type 2 Diabetic Patients Inadequately Controlled With Metformin Plus Sulphonylurea.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC20965; 2008-001855-23
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin; taspoglutide

ARMS (3):
- insulin glargine (Active Comparator): insulin glargine starting dose 10 IU daily in addition to continued prestudy metformin treatment
  Interventions: Drug: insulin glargine; Drug: metformin
- taspoglutide 10 mg (Experimental): taspoglutide 10 mg once weekly in addition to continued prestudy metformin treatment
  Interventions: Drug: metformin; Drug: taspoglutide
- taspoglutide 10 mg/20 mg (Experimental): taspoglutide 20 mg once weekly (after 4 weeks of taspoglutide 10 mg once weekly) in addition to continued prestudy metformin treatment
  Interventions: Drug: metformin; Drug: taspoglutide

INTERVENTIONS:
Drug: insulin glargine — starting dose 10 IU daily
  Arms: insulin glargine
Drug: metformin — As prescribed
Drug: taspoglutide — 10 mg once weekly
  Arms: taspoglutide 10 mg
Drug: taspoglutide — 20 mg once weekly (after 4 weeks of taspoglutide 10 mg once weekly)
  Arms: taspoglutide 10 mg/20 mg

SUMMARY:
This 3-arm study will assess the efficacy, safety and tolerability of taspoglutide compared to insulin glargine in patients with insulin-naive type 2 diabetes mellitus inadequately controlled with metformin and sulphonylurea combination therapy. Patients will be randomized to receive taspoglutide (10 mg once weekly, or 10mg once weekly for 4 weeks followed by 20mg once weekly) or insulin glargine (starting dose 10 IU/day) in a ratio of 1:1:1 in addition to continued prestudy metformin treatment. The anticipated time on study treatment is 2+ years, and the target sample size if 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes treated with a stable dose of metformin and sulphonylurea for at least 12 weeks;
* C-peptide (fasting) >=1.0ng/mL;
* HbA1c >=7.0% and <=10.0% at screening;
* BMI >=25 (>23 for Asians) and <=45kg/m2 at screening;
* stable weight +-5% for at least 12 weeks prior to screening.

Exclusion Criteria:

* history of type 1 diabetes mellitus or acute metabolic diabetic complications such as ketoacidosis or hyperosmolar coma in the previous 6 months;
* evidence of clinically significant diabetic complications;
* symptomatic poorly controlled diabetes;
* clinically symptomatic gastrointestinal disease;
* myocardial infarction, coronary artery bypass surgery, post-transplantation cardiomyopathy or stroke within the previous 6 months;
* known hemoglobinopathy or chronic anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose; change from baseline in body weight; responder rates for HbA1c (target <=7.0%, <=6.5%); incidence of hypoglycemia; change from baseline in lipid profile. | 24 weeks
Relative change in glucose, insulin, C-peptide and glucagon during a meal tolerance test. | 24 weeks
Safety: Adverse events, vital signs, physical examination, clinical laboratory tests, ECG and anti-taspoglutide antibodies | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (184):
- United States (66):
  - Phoenix, Arizona
  - Searcy, Arkansas
  - Concord, California
  - Huntington Beach, California
  - Los Angeles, California
  - Los Gatos, California
  - Roseville, California
  - San Diego, California
  - Santa Ana, California
  - Westlake Village, California
  - Washington D.C., District of Columbia
  - Green Cove Springs, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Ormond Beach, Florida
  - Oviedo, Florida
  - Palm Harbor, Florida
  - Trinity, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Quincy, Illinois
  - Springfield, Illinois
  - Avon, Indiana
  - Indianapolis, Indiana
  - Arkansas City, Kansas
  - Crestview Hills, Kentucky
  - Metairie, Louisiana
  - Sunset, Louisiana
  - Portland, Maine
  - North East, Maryland
  - Worchester, Massachusetts
  - Saint Claire Shores, Michigan
  - Jackson, Mississippi
  - Picayune, Mississippi
  - Springfield, Missouri
  - Grand Island, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Blackwood, New Jersey
  - Cherry Hill, New Jersey
  - Moorestown, New Jersey
  - Toms River, New Jersey
  - Albany, New York
  - Flushing, New York
  - Mineola, New York
  - Asheville, North Carolina
  - Harrisburg, North Carolina
  - Fargo, North Dakota
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Genoa, Ohio
  - Toledo, Ohio
  - Altoona, Pennsylvania
  - Bensalem, Pennsylvania
  - Feasterville, Pennsylvania
  - Harrisburg, Pennsylvania
  - Jefferson Hills, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Tipton, Pennsylvania
  - Orangeburg, South Carolina
  - Johnson City, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Waukesha, Wisconsin
- Australia (3):
  - St Leonards, New South Wales
  - Wollongong, New South Wales
  - Freemantle, Queensland
- Austria (3):
  - Graz
  - Salzburg
  - Vienna
- Belgium (4):
  - Arlon
  - Bonheiden
  - Leuven
  - Liège
- Brazil (5):
  - Campina Grande do Sul, Paraná
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (6):
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Pointe-Claire, Quebec
  - Sherbrooke, Quebec
- Czechia (5):
  - Brno
  - Havířov
  - Pilsen
  - Prague
  - Trutnov
- Finland (3):
  - Helsinki
  - Jyväskylä
  - Tampere
- France (12):
  - Avignon
  - Besançon
  - Bois-Guillaume
  - Brest
  - Corbeil-Essonnes
  - La Rochelle
  - Marseille
  - Montpellier
  - Nîmes
  - Paris
  - Strasbourg
  - Vénissieux
- Germany (11):
  - Bad Lauterberg im Harz
  - Berlin
  - Bochum
  - Bosenheim
  - Dortmund
  - Falkensee
  - Freiburg im Breisgau
  - Mainz
  - Offenbach a.M.
  - Reichenbach
  - Würzburg
- Greece (3):
  - Athens
  - Larissa
  - Thessaloniki
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Hungary (3):
  - Balatonfüred
  - Budapest
  - Szekszárd
- Italy (5):
  - Napoli, Campania
  - Rome, Lazio
  - Codogno, Lombardy
  - Milan, Lombardy
  - Turin, Piedmont
- Mexico (4):
  - Aguascalientes
  - Cuernavaca
  - Monterrey
  - Tampico
- Auckland, New Zealand
- Peru (3):
  - Arequipa
  - Lima
  - Trujillo
- Poland (7):
  - Grodzisk Mazowiecki
  - Kamieniec Ząbkowicki
  - Lodz
  - Rzeszów
  - Sobótka
  - Szczecin
  - Wroclaw
- Portugal (2):
  - Coimbra
  - Lisbon
- Puerto Rico (6):
  - Guyanabo, San Juan
  - Levittown
  - Orocovis
  - Ponce
  - San Juan
  - Trujillo Alto
- Russia (8):
  - Barnaul
  - Chelyabinsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Tomsk
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- South Korea (3):
  - Daegu
  - Incheon
  - Seoul
- Spain (8):
  - Almería, Almeria
  - Barcelona, Barcelona
  - Granada, Granada
  - Pozuelo de Alarcón, Madrid
  - Seville, Sevilla
  - Alzira, Valencia
  - Valencia, Valencia
  - Valladolid, Valladolid
- Bangkok, Thailand
- United Kingdom (6):
  - Atherstone
  - Chesterfield
  - Dumfries
  - Liverpool
  - Sheffield
  - Trowbridge

REFERENCES:
- [Derived] Nauck M, Horton E, Andjelkovic M, Ampudia-Blasco FJ, Parusel CT, Boldrin M, Balena R; T-emerge 5 Study Group. Taspoglutide, a once-weekly glucagon-like peptide 1 analogue, vs. insulin glargine titrated to target in patients with Type 2 diabetes: an open-label randomized trial. Diabet Med. 2013 Jan;30(1):109-13. doi: 10.1111/dme.12003. PMID 22937895